CLINICAL TRIAL: NCT07106970
Title: Linear Ablation Added to Pulmonary Vein Isolation Versus Pulmonary Vein Isolation Alone Using Pulsed Field Ablation for Persistent Atrial Fibrillation: a Multi-center Randomized Controlled Trial
Brief Title: PVI Alone vs PVI and Linear Ablation for Persistent Atrial Fibrillation (PROMPT AF II)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PF336
Record Dates: First submitted 2025-07-23; First posted 2025-08-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicenter, open-label, randomized controlled trial to investigate whether a linear ablation in addition to pulmonary vein isolation (PVI) outperforms PVI alone using pulsed field ablation (PFA) in maintaining sinus rhythm for persistent atrial fibrillation (PerAF)
Who Masked: Participant, Investigator
Masking Description: The control group will consist of subjects randomized into PVI alone arm, who will accept bilateral PVI only with the same study device as those used in the Test group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI and linear ablation arm (Experimental): Subjects in PVI and linear ablation arm will undergo bilateral PVI, and linear ablations in the posterior wall (PW), mitral isthmus (MI) and cavo-tricuspid isthmus (CTI) using the study device, and EIVOM could be performed additionally before or after PFA at the operator's discretion.
  Interventions: Procedure: Linear ablation; Procedure: PVI alone
- PVI alone arm (Active Comparator): Subjects randomized to the PVI alone arm will undergo PVI only with the study device.
  Interventions: Procedure: PVI alone

INTERVENTIONS:
Procedure: Linear ablation — Linear ablations in the posterior wall (PW), mitral isthmus (MI) and cavo-tricuspid isthmus (CTI) using the study device.EIVOM could be performed additionally before or after PFA at the operator's discretion.
  Arms: PVI and linear ablation arm
Procedure: PVI alone — Undergo PVI with the study device

SUMMARY:
This study is a prospective, multicenter, open-label, randomized controlled trial to investigate whether a linear ablation in addition to pulmonary vein isolation (PVI) outperforms PVI alone using pulsed field ablation (PFA) in maintaining sinus rhythm for persistent atrial fibrillation (PerAF)

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, randomized controlled trial to investigate whether a linear ablation in addition to PVI outperforms PVI alone using PFA in maintaining sinus rhythm for PerAF. Enrolled subjects will be randomized by the ratio of 1:1 into PVI and linear ablation arm or PVI alone arm. Subjects in PVI and linear ablation arm will undergo bilateral PVI, and linear ablations in the posterior wall (PW), mitral isthmus (MI) and cavo-tricuspid isthmus (CTI) using the study device and EIVOM could be performed additionally before or after PFA at the operator's discretion, it is recommended to perform EIVOM first. Subjects randomized to the PVI alone arm will undergo PVI only. If atrial fibrillation (AF) cannot be terminated during ablation, cardioversion will be performed. After ablation, all the subjects will be followed at discharge, 1 month and then at 3-month intervals up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

Study subjects are required to meet all the following inclusion criteria:

1. Subjects with an age range of 18 years or above and 80 years or below.
2. Subjects have symptomatic, drug-resistant, persistent AF, defined as:

   1. Symptomatic: these symptoms include but not limited to palpitations, presyncope, syncope, fatigue, and shortness of breath.
   2. Drug-resistant: effectiveness failure of, intolerance to, or specific contraindication to at least one AAD.
   3. Persistent: continuous AF for > 90 days, i) with a minimum a physician's note confirming the diagnosis AND,within 180 days of Enrollment Date, either a 24-hour or longer continuous ECG recording confirming continuous AF OR Two ECGs showing continuous AF taken at least 90 days apart.
3. Subjects undergoing a first-time ablation procedure for AF.
4. Subjects who are willing and capable of providing ICF and participating in all testing associated with this study.

Exclusion Criteria:

1. AF that is secondary to electrolyte imbalance, thyroid disease, alcohol, or other reversible/non-cardiac causes.
2. Left atrial anteroposterior diameter ≥ 6.0 cm by transthoracic echocardiography (TTE) within 3 months prior the procedure.
3. Heart failure with left ventricular ejection fraction (LVEF) < 30% by TTE within 3 months prior the procedure.
4. LA thrombus detected by Transesophageal Echocardiography (TEE) or cardiac CT within one day before the procedure or Intracardiac Echocardiography (ICE) before atrial septal puncture during the procedure.
5. Current or anticipated pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices, mechanical valve, interatrial baffle, closure device, patch, or patent foramen oval occlude, left atrial appendage closure at the time of ablation.
6. Any of the following events within 90 days of the Consent Date:

   1. Myocardial infarction, unstable angina or coronary intervention or any cardiac surgery
   2. Pericarditis or symptomatic pericardial effusion
   3. Gastrointestinal bleeding
   4. Stroke, transient ischemic attack (TIA), or intracranial bleeding or any non-neurologic thromboembolic event
7. Contraindication to, or unwillingness to use systemic anticoagulation.
8. Subjects cannot be removed from Class I/III AAD for reasons other than atrial arrhythmia.
9. Women of childbearing potential who are pregnant or lactating.
10. Renal insufficiency if an estimated glomerular filtration rate (eGFR) is < 30 mL/min/1.73 m2, or with any history of renal dialysis or renal transplant.
11. Conditions that in the investigator's medical opinion would interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation.
12. Predicted life expectancy less than 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint with Treatment Success. | Completion of treatment 360 days compared with the baseline
  Number of Participants free from Arrhythmia, Re-ablation, Cardioversion, and AAD use.
Primary Safety Endpoint with Safety events related to AF catheter ablation. | Completion of treatment 360 days compared with the baseline
  Number of Participants with following device or procedure-related serious Composite Adverse Events (CAEs).

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoint with Chronic Success. | Completion of treatment 360 days compared with the baseline.
  Number of Participants with Chronic Success, Freedom from any documented AF, AFL or AT episode lasting ≥10s via 12-lead ECG or ≥30s via Holter (or other continuous rhythm monitoring device) on/off AADs after the blanking period to Day 360.
Secondary Safety Endpoint with Non-SAE. | Completion of treatment 360 days compared with the baseline
  Number of Participants with Non-Serious Composite Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Doctor, Principal Investigator — Beijing Anzhen Hospital of the Capital University of Medical Sciences
Locations (1):
- Beijing Anzhen Hospital, affiliated to Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No